CLINICAL TRIAL: NCT01659749
Title: Educational, Social Support, and Nutritional Interventions and Their Cumulative Effect on Pregnancy Outcomes and Quality of Life in Teen and Adult Women With Phenylketonuria (PKU) or Maple Syrup Urine Disease (MSUD).
Brief Title: Educational, Social Support, and Nutritional Interventions and Their Cumulative Effect on Pregnancy Outcomes and Quality of Life in Teen and Adult Women With Phenylketonuria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rani Singh, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00002447a
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy; Phenylketonuria
Keywords: Genetics; Metabolic; Nutrition; Maternal PKU; Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias; Phenylketonuria, Maternal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic Camp (Other): Metabolic Camp is an educational and social support program for females age 11 through adult with phenylketonuria (PKU) and maple syrup urine disease (MSUD), two inherited metabolic disorders (IMD). Camp provides a supportive environment for adolescent girls and women to learn about the importance of nutrition and diet self-management, with the intention of arresting the disease process and minimizing the instances of miscarriages and severe birth defects, which are high in this population. After 20+ years, Metabolic Camp is established as a unique, national program allowing up to 35 campers to live and learn during a week of nutritional support and productive activities, while simultaneously providing researchers an opportunity to gather important data.
  Interventions: Behavioral: Metabolic camp

INTERVENTIONS:
Behavioral: Metabolic camp — To use an recreational camp setting to instruct PKU females of reproductive age how to make responsible dietary and reproductive decisions.

SUMMARY:
The purpose of this project is to study the effectiveness of teaching teens and young women with Phenylketonuria (PKU) or Maple Syrup Urine Disease (MSUD) about their disease and nutrition related issues in a camp environment. It will also look at pregnancy outcome results in women with PKU who attended Metabolic Camp and compare their results to other women with PKU who have not attended the Metabolic Camp.

DETAILED DESCRIPTION:
Metabolic Camp is an educational and social support program with research opportunities that was developed in 1995 by Rani H. Singh, PhD, RD for females age 11 through adult with phenylketonuria (PKU) and maple syrup urine disease (MSUD), two inherited metabolic disorders (IMD). Camp provides a supportive environment for adolescent girls and women to learn about the importance of nutrition and diet self-management, with the intention of arresting the disease process and minimizing the instances of miscarriages and severe birth defects, which are high in this population. After 20+ years, Metabolic Camp is established as a unique, national program allowing up to 35 campers to live and learn during a week of nutritional support and productive activities, while simultaneously providing researchers an opportunity to gather important data.

The aims of Metabolic Camp are 1) to implement education curriculum and support activities as an intervention program for females with PKU and MSUD, 2) to evaluate knowledge of disease and dietary management, dietary treatment compliance, quality of life, and reproductive choice issues and assess change in outcomes post-Camp, 3) to gather data through the implementation of a research protocol during baseline and post-Camp each year, and 4) to provide clinical and research training in IMD for professionals, from dietitians to medical students. Campers must complete an informed consent process, should they decide to participate in research activities. All campers submit a three-day food record and blood samples to measure plasma amino acids on the first and last day of camp, both of which are not classified as research activities, but rather standard of care for their disorder. Additional studies such as indirect calorimetry, bone health markers, anthropometric markers, nutritional status, mental and emotional wellbeing, neurocognitive functioning, access to disease specific care, metabolomic profiling, gut microbiota, and blood and urine analysis, have been and may continue to be assessed in those who participate in research pre and post-Camp. These are novel investigations for the study of IMD and essential to understand the physiological effects of Camp.

In over 20 years of Metabolic Camp, the following data have been collected: health history and demographics, anthropometrics, dietary intake, compliance with medically prescribed diet, quality of life, physical activity, plasma amino acids, select blood and urine biomarkers, and bone density. Data are stored in REDCap, allowing evaluation of short- and long-term outcomes on the life course of females with PKU and MSUD. Each year, phenylalanine (Phe)/leucine (Leu) blood concentrations of campers decrease over the one week camp period, demonstrating better metabolic control and compliance with diet. Campers' knowledge of disease etiology, management, and effects, including Maternal PKU Syndrome (MPKU) are improved. Social support networks are strengthened by meeting peers with the same or similar disorder. The study protocol includes a comprehensive assessment of blood and urine biomarkers to examine PKU from a much broader approach compared to the traditional measurement of a single biomarker to assess patient status. Beneficial to campers and clinicians alike, Metabolic Camp is an invaluable experience to gain insight, knowledge, and stimulate new ideas related to research and optimal patient care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PKU or other aminoacidopathy, female, age 11 or older, able to provide informed consent

Exclusion Criteria:

* Those not fitting the inclusion criteria

Inclusion Criteria for healthy controls

Individuals eligible to participate in this study must meet all of the following criteria:

* Adult camp counselors or staff determined to be in good health.
* Not diagnosed with PKU, MSUD or other hereditary metabolic disorder
* Willing and able to provide written informed consent
* Willing and able to comply with relevant camp guidelines and study procedures

Min Age: 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1995-06 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2037-07 (Estimated)

PRIMARY OUTCOMES:
Change in plasma Amino Acid concentration | Baseline, Week 1
  Concentration of Phenylalanine in plasma (measured in mg/dL) will be measured the first day of metabolic camp and at the last day of the camp.
Change in Dietary intake of Phenylalanine | Baseline, Week 1
  Dietary intake of Phenylalanine (measured in mg/Kg) will be measured the first day of metabolic camp and at the last day of the camp, using a three-day diet food record that has been completed at baseline and post-camp.

CONTACTS AND LOCATIONS:
Overall Officials: Rani H Singh, PhD RD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Human Genetics, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jani R, Coakley K, Douglas T, Singh R. Protein intake and physical activity are associated with body composition in individuals with phenylalanine hydroxylase deficiency. Mol Genet Metab. 2017 Jun;121(2):104-110. doi: 10.1016/j.ymgme.2017.04.012. Epub 2017 Apr 28. PMID 28465125

DOCUMENTS (2):
  • Informed Consent Form: assent form (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT01659749/ICF_000.pdf
  • Informed Consent Form: assent Form (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT01659749/ICF_001.pdf